CLINICAL TRIAL: NCT00748969
Title: Phase II/III, Randomized, Clinical Trial of the Effects of Nutropin AQ® on Growth and Bone Metabolism in Children With MPS I, II, and VI and Short Stature
Brief Title: Clinical Trial of Growth Hormone in MPS I, II, and VI
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Insufficient recruitment.
Sponsor: Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0808M43681
Record Dates: First submitted 2008-09-08; First posted 2008-09-09 (Estimated); Results first posted 2014-11-24 (Estimated); Last update posted 2018-09-05 (Actual); Status verified 2014-11

CONDITIONS: Mucopolysaccharidosis I; Mucopolysaccharidosis II; Mucopolysaccharidosis VI
Keywords: MPS I; MPS II; MPS VI; growth hormone; short stature
MeSH Terms: conditions — Mucopolysaccharidosis I; Mucopolysaccharidosis II; Mucopolysaccharidosis VI; Sudden Infant Death; Dwarfism | interventions — Human Growth Hormone; Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Growth hormone treatmen (Experimental): Growth hormone treatment arm. Somatropin (DNA origin)
  Interventions: Drug: Somatropin (DNA origin)
- No growth hormone treatment in year 1 (No Intervention): No growth hormone treatment in year 1; option for treatment in year 2 open-label period.

INTERVENTIONS:
Drug: Somatropin (DNA origin) — The study starting dose of Nutropin AQ® will be 0.48 mg/kg/week divided into daily SC injections. Nutropin AQ® will be administered by either the subject or, if unable to demonstrate competency in this, then by the guardian. To decrease the risk of increased intracranial hypertension, the dose in the first month of treatment will be decreased by 50% (0.24 mg/kg/week), and then increased to 0.48 mg/kg/week if tolerated well after 1 month.
  Other Names: Nutropin AQ
  Arms: Growth hormone treatmen

SUMMARY:
The purpose of this study is to determine whether growth hormone is a safe and effective treatment for short stature in children with Mucopolysaccharidosis type I, II, and VI.

DETAILED DESCRIPTION:
Although children with MPS I, II, and VI who are treated with Hematopoietic Cell Transplantation (HCT) and/or enzyme replacement therapy (ERT) are living into adulthood with good cognitive development, their quality of life is significantly impacted by their skeletal abnormalities (i.e., kyphosis, scoliosis, and genu valgum), contractures, and severe short stature. Here at the University of Minnesota we have seen some promising clinical outcomes in children with MPS IH whom we have treated with human growth hormone (hGH). There are currently no reports in the literature of the impact of treating children with MPS and short stature, with hGH on their growth velocity or characteristic skeletal abnormalities. This study will advance the care of these children by providing data in this yet unexplored area of pediatric medicine with the goal of improving the quality of life for these children by improving height, mobility, and neuropsychological functioning.

This is a Phase II/III randomized, single-center, 12 month clinical trial of growth hormone in male and female participants with MPS I, II, or VI, followed by 12 months open label. Participants with height ≤ -2 SDS for age and gender will be randomized for the first 12 months 1:1 to treatment or no treatment. At the conclusion of the 12 months, all subjects will be offered an additional 12 months of treatment.

ELIGIBILITY:
Inclusion Criteria:

* A parent or legally authorized representative must provide written informed consent and comply with study assessments for the full duration of the study.
* Chronologic age ≥ 5 years and bone age ≤12 years
* Diagnosis of MPS I, II, or VI
* Height ≤ -2 SDS for age and gender
* Ability to travel to study center for evaluations.
* Ability of the participant to cooperate with study procedures, to notify a guardian of symptoms, and provide assent for participation in the study.

Exclusion Criteria:

* History of treatment with hGH
* Untreated pituitary deficiency
* Pregnancy (positive urine pregnancy test) prior to enrollment in the study
* Participation in another simultaneous medical intervention trial
* Patients with closed epiphysis
* Active neoplasm
* Orthopedic procedure of the femur within the last 6 months.
* Known or suspected allergy to trial product or related products.
* Structural lesion on brain MRI resulting in brain compression
* Any other social or medical condition that the investigator believes would pose a significant hazard to the subject if the investigational therapy were initiated or be detrimental to the study.
* Obstructive sleep apnea without BiPAP or tonsillectomy/adenoidectomy treatment.
* CNS shunt.
* Abnormal cardiac function based on echocardiogram within 6 months prior to enrollment :
* Ejection fraction less than 50%
* Left ventricular chamber size greater than or less than 2 standard deviations of normal for body surface area
* Left ventricular wall thickness greater than or less than 2 standard deviations of normal for body surface area
* More than mild to moderate aortic insufficiency with abdominal aortic run-off
* More than mild to moderate mitral insufficiency with pulmonary hypertension
* Abnormal pulmonary function based on pulmonary function tests within 6 months prior to enrollment:
* abnormal FVC < 80% of predicted for age, gender, and height
* abnormal FEV1 < 80% predicted for age, gender, and height
* abnormal FEV1/FVC
* abnormal oxygen saturation

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2 (Actual)
Dates: Start 2008-11; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lynda E Polgreen, M.D., Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Growth Hormone Treatmen | No Growth Hormone Treatment in Year 1
Started | 1 (Subject withdrew from study due to worsening sleep apnea) | 1 (Subject withdrew from study due to randomization to no treatment)
Completed | 0 | 0
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Growth Hormone Treatmen | No Growth Hormone Treatment in Year 1 | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Continuous [Mean (Full Range); unit: years] | 10.9 [10.9 to 10.9] | 13.5 [13.5 to 13.5] | 12.2 [10.9 to 13.5]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 1 | 2
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in Growth Velocity From Baseline to End of Study Year 1.
Time Frame: 12 months
Population: Zero participants analyzed in the "No growth hormone treatment" group due to subject withdrew from study as soon as informed they were assigned the no treatment group.
Measure: Number; unit: cm/yr
Groups:
- Growth Hormone Treatment: Growth hormone treatment arm. Somatropin (DNA origin)
  Somatropin (DNA origin): The study starting dose of Nutropin AQ® will be 0.48 mg/kg/week divided into daily SC injections. Nutropin AQ® will be administered by either the subject or, if unable to demonstrate competency in this, then by the guardian. To decrease the risk of increased intracranial hypertension, the dose in the first month of treatment will be decreased by 50% (0.24 mg/kg/week), and then increased to 0.48 mg/kg/week if tolerated well after 1 month.
- No Growth Hormone Treatment: Observation only: no growth hormone treatment and no placebo.
Arm/Group | Growth Hormone Treatment | No Growth Hormone Treatment
Number analyzed (Participants) | 1 | 0
cm/yr | NA — insufficient data due to study termination |

2. Secondary Outcome: Safety: Number Drug Related SAEs
Time Frame: 1 months
Population: Study stopped early due to inability to enroll participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Growth Hormone Treatment | No Growth Hormone Treatment
Number analyzed (Participants) | 1 | 0
Participants | 0 | 0

ADVERSE EVENTS:
Description: Zero participants analyzed in the "No growth hormone treatment" group due to subject withdrew from study as soon as informed they were assigned the no treatment group.
Groups:
- GH Treatment: Growth hormone treatment arm. Somatropin (DNA origin)
  Somatropin (DNA origin): The study starting dose of Nutropin AQ® will be 0.48 mg/kg/week divided into daily SC injections. Nutropin AQ® will be administered by either the subject or, if unable to demonstrate competency in this, then by the guardian. To decrease the risk of increased intracranial hypertension, the dose in the first month of treatment will be decreased by 50% (0.24 mg/kg/week), and then increased to 0.48 mg/kg/week if tolerated well after 1 month.
- No GH Treatment: No placebo/no treatment
Arm/Group | GH Treatment | No GH Treatment
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 1/1 | 0/0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GH Treatment (N=1) | No GH Treatment (N=0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
worsening OSA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes